CLINICAL TRIAL: NCT02805660
Title: A Phase 1/2 Study of HDAC Inhibitor, Mocetinostat, in Combination With PD-L1 Inhibitor, Durvalumab, in Advanced or Metastatic Solid Tumors and Non-Small Cell Lung Cancer
Brief Title: Phase 1/2 Study of Mocetinostat and Durvalumab in Patients With Advanced Solid Tumors and NSCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was discontinued early because the Sponsor de-prioritized development of mocetinostat. The decision to stop was not due to any patient safety issues.
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0103-020
Record Dates: First submitted 2016-06-10; First posted 2016-06-20 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Advanced Cancer
Keywords: MGCD0103; MEDI4736; Mocetinostat; Durvalumab; HDAC Inhibitor; PD-L1 Inhibitor; Phase 1; Phase 2; Metastatic Solid Tumor; Non-small cell lung cancer; immunotherapy; checkpoint inhibitor
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — mocetinostat; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Phase 1: Dose Escalation - 50 mg (Experimental): The Phase 1 dose escalation established the recommended phase 2 dose (RP2D) of mocetinostat. Participants with advanced solid tumors were included in this Phase.
  Interventions: Drug: Mocetinostat - 50 mg; Drug: Durvalumab - 1500 mg
- Phase 1: Dose Escalation - 70 mg (Experimental): The Phase 1 dose escalation established the recommended phase 2 dose (RP2D) of mocetinostat. Participants with advanced solid tumors were included in this Phase.
  Interventions: Drug: Mocetinostat - 70 mg; Drug: Durvalumab - 1500 mg
- Phase 1: Dose Escalation - 90 mg (Experimental): The Phase 1 dose escalation established the recommended phase 2 dose (RP2D) of mocetinostat. Participants with advanced solid tumors were included in this Phase.
  Interventions: Drug: Mocetinostat - 90 mg; Drug: Durvalumab - 1500 mg
- Phase 2: Combination Regimen - Cohort 1 (Experimental): Participants with non-small cell lung cancer (NSCLC) who were naïve to treatment with immunotherapy, and had a tumor with no/low programmed cell death ligand 1 (PD-L1) expression were included in this cohort.
  Interventions: Drug: Mocetinostat - Recommended Phase 2 Dose (70 mg); Drug: Durvalumab - 1500 mg
- Phase 2: Combination Regimen - Cohort 2 (Experimental): Participants with non-small cell lung cancer (NSCLC) who were naïve to treatment with immunotherapy, and had a tumor with high programmed cell death ligand 1 (PD-L1) expression were included in this cohort.
  Interventions: Drug: Mocetinostat - Recommended Phase 2 Dose (70 mg); Drug: Durvalumab - 1500 mg
- Phase 2: Combination Regimen - Cohort 3 (Experimental): Participants with non-small cell lung cancer (NSCLC) who have been previously treated with an anti-programmed cell death ligand 1 (PD-L1) or anti-programmed cell death 1 (PD-1) agent with clinical benefit response followed by progression of disease were included in this cohort.
  Interventions: Drug: Mocetinostat - Recommended Phase 2 Dose (70 mg); Drug: Durvalumab - 1500 mg
- Phase 2: Combination Regimen - Cohort 4 (Experimental): Participants with non-small cell lung cancer (NSCLC) who have been previously treated with an anti-programmed cell death ligand 1 (PD-L1) or anti-programmed cell death 1 (PD-1) agent who had progression of disease ≤ 16 weeks after initiation of treatment were included in this cohort.
  Interventions: Drug: Mocetinostat - Recommended Phase 2 Dose (70 mg); Drug: Durvalumab - 1500 mg

INTERVENTIONS:
Drug: Mocetinostat - 50 mg — Participants received mocetinostat three times weekly as an oral capsule.
  Other Names: MGCD0103
  Arms: Phase 1: Dose Escalation - 50 mg
Drug: Mocetinostat - 70 mg — Participants received mocetinostat three times weekly as an oral capsule.
  Other Names: MGCD0103
  Arms: Phase 1: Dose Escalation - 70 mg
Drug: Mocetinostat - 90 mg — Participants received mocetinostat three times weekly as an oral capsule.
  Other Names: MGCD0103
  Arms: Phase 1: Dose Escalation - 90 mg
Drug: Mocetinostat - Recommended Phase 2 Dose (70 mg) — Participants received mocetinostat three times weekly as an oral capsule, at the dose recommended after Phase 1 (70 mg).
  Other Names: MGCD0103
  Arms: Phase 2: Combination Regimen - Cohort 1; Phase 2: Combination Regimen - Cohort 2; Phase 2: Combination Regimen - Cohort 3; Phase 2: Combination Regimen - Cohort 4
Drug: Durvalumab - 1500 mg — Participants received durvalumab as an intravenous infusion every 4 weeks.
  Other Names: MEDI4736

SUMMARY:
Mocetinostat (MGCD0103) is an orally administered HDAC inhibitor. Durvalumab (MEDI4736) is a human monoclonal antibody that is an inhibitor of the Programmed Cell Death Ligand (or PD-L1). Durvalumab is also known as a checkpoint inhibitor.

This study is evaluating the combination regimen of mocetinostat and durvalumab in participants with Advanced or Metastatic Solid Tumors and Non-Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1-Diagnosis of advanced or metastatic solid tumor; Phase 2-Diagnosis of NSCLC
* Not amenable to treatment with curative intent
* Adequate bone marrow and organ function

Exclusion Criteria:

* Impaired heart function
* Uncontrolled tumor in the brain
* Other active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Southern Cancer Center, PC, Mobile, Alabama
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Woodlands Medical Specialists - Pensacola, Pensacola, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Unniversity of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Shenandoah Oncology - Winchester, Winchester, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2: Combination Regimen - Cohort 1: Participants with non-small cell lung cancer (NSCLC) who were naïve to treatment with immunotherapy, and had a tumor with no/low programmed cell death ligand 1 (PD-L1) expression were included in this cohort.
  Durvalumab - 1500 mg: Participants received durvalumab as an intravenous infusion every 4 weeks.
  Mocetinostat - Recommended Phase 2 Dose (70 mg): Participants received mocetinostat three times weekly as an oral capsule, at the dose recommended after Phase 1 (70mg).
- Phase 2: Combination Regimen - Cohort 2: Participants with non-small cell lung cancer (NSCLC) who were naïve to treatment with immunotherapy, and had a tumor with high programmed cell death ligand 1 (PD-L1) expression were included in this cohort.
  Durvalumab - 1500 mg: Participants received durvalumab as an intravenous infusion.
  Mocetinostat - Recommended Phase 2 Dose (70 mg): Participants received mocetinostat three times weekly as an oral capsule, at the dose recommended after Phase 1 (70 mg).
Period: Overall Study
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
Started | 5 | 4 | 11 | 18 | 3 | 23 | 19
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 4 | 11 | 18 | 3 | 23 | 19
Not completed — Death | 5 | 2 | 9 | 5 | 0 | 14 | 12
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 1 | 0 | 2
Not completed — Study terminated by Sponsor | 0 | 0 | 1 | 4 | 2 | 3 | 1
Not completed — Miscellaneous | 0 | 1 | 0 | 4 | 0 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4 | Total
Number analyzed (Participants) | 5 | 4 | 11 | 18 | 3 | 23 | 19 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 4 | 5 | 0 | 9 | 9 | 33
  >=65 years | 2 | 1 | 7 | 13 | 3 | 14 | 10 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6 | 12 | 1 | 9 | 8 | 42
  Male | 1 | 2 | 5 | 6 | 2 | 14 | 11 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 7
  Not Hispanic or Latino | 5 | 3 | 10 | 17 | 2 | 20 | 19 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 5
  White | 5 | 3 | 8 | 14 | 3 | 18 | 16 | 67
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 11 | 18 | 3 | 23 | 19 | 83
Smoking History [Count of Participants; unit: Participants]
  Non-smoker | 4 | 3 | 6 | 3 | 0 | 3 | 2 | 21
  Current Smoker | 1 | 1 | 0 | 3 | 0 | 3 | 2 | 10
  Former Smoker | 0 | 0 | 5 | 12 | 3 | 17 | 15 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience a Dose-Limiting Toxicity (DLT) During the First 28-day Cycle of Combination Treatment In Phase 1
Description: Toxicities were graded using the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03. Any of the following events considered to be causally related to treatment with mocetinostat in combination with durvalumab that occurred during Phase 1 were considered a DLT:
  * Any Grade 4 immune-related adverse event (irAE)
  * Grade 3 or greater colitis
  * Grade 3 or greater noninfectious pneumonitis
  * Grade 2 pneumonitis that did not resolve to ≤ Grade 1 within 3 days of the initiation of maximal supportive care
  * Grade 3 irAE (excluding colitis or pneumonitis) that:
    * Did not resolve to Grade 2 within 3 days after onset of the event despite optimal medical management including systemic corticosteroids, or
    * Did not resolve to Grade ≤1 or Baseline within 14 days
  * Liver transaminase elevation >8×upper limit of normal (ULN) or total bilirubin >5×ULN
  * Grade 3 or greater non-irAE, except nausea, vomiting, anorexia, dehydration, or diarrhea
Time Frame: 28 days
Population: DLT Evaluable Population - Participant must have either been on study for one full cycle and have received treatment with durvalumab and at least 9 of 12 scheduled mocetinostat doses (75%) in Cycle 1 or have experienced a DLT in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg
Number analyzed (Participants) | 4 | 3 | 6
Participants | 0 | 0 | 0

2. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) was defined as the number of participants documented to have a confirmed Complete Response (CR) or Partial Response (PR). Complete Response was defined as the complete disappearance of all target lesions with the exception of nodal disease. Partial Response was defined at least a 30% decrease in the sum of diameters of target measurable lesions. Responses were determined by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Participants without response data were counted as non-responders.
  Inferential statistical analyses were conducted for Phase 2 only, as efficacy was not part of the Phase 1 objectives.
Time Frame: Up to approximately 10 months
Population: Clinical Activity Evaluable Population - The Clinical Activity Evaluable Population was defined as all participants who had at least one on-study disease assessment or discontinued from treatment for progressive disease (PD).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
Number analyzed (Participants) | 5 | 4 | 9 | 15 | 3 | 21 | 13
Percentage of participants | 0 [0.0 to 52.2] | 0 [0.0 to 60.2] | 0 [0.0 to 33.6] | 6.7 [0.2 to 31.9] | 0 [0.0 to 70.8] | 9.5 [1.2 to 30.4] | 23.1 [5.0 to 53.8]
Statistical Analysis 1: Comparison: Phase 2: Combination Regimen - Cohort 1; Test type: Superiority — An exact test for single proportion was performed to test null hypothesis (H0): ORR <= 5% against alternative hypothesis (H1): ORR > 5% for Cohorts 1, 3, and 4 and to test H0: ORR <= 27% against H1: ORR > 27% for Cohort 2; p = 0.537, Exact Test
Statistical Analysis 2: Comparison: Phase 2: Combination Regimen - Cohort 2; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p > 0.999, Exact Test
Statistical Analysis 3: Comparison: Phase 2: Combination Regimen - Cohort 3; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.283, Exact Test
Statistical Analysis 4: Comparison: Phase 2: Combination Regimen - Cohort 4; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.025, Exact Test

3. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events
Time Frame: Day 1 to 28 days after last dose of study treatment (up to a maximum of 125 weeks in phase 1 and a maximum of 92 weeks in phase 2)
Population: Safety Population - The Safety population was defined as all participants who received at least 1 dose of either mocetinostat or durvalumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
Number analyzed (Participants) | 5 | 4 | 11 | 18 | 3 | 23 | 19
Participants | 5 | 4 | 10 | 18 | 3 | 23 | 18

4. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time in days from date of the first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the first documentation of objective Progressive Disease (PD) or to death due to any cause in the absence of documented PD. DR was only calculated for the subgroup of participants who achieved a Best Overall Response of CR or PR and was presented for responses assessed by Investigator's assessment.
  Data is displayed for Phase 2 only, as no participants experienced an objective response (CR or PR) during Phase 1.
Time Frame: Up to approximately 10 months
Population: Clinical Activity Evaluable Population (Subgroup of Responders) - Duration of response was only calculated for the subgroup of participants achieving a CR or PR.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
Number analyzed (Participants) | 1 | 0 | 2 | 3
Days | 115 [NA to NA] — Due to a small number of participants and events, data was not estimable. |  | 329 [NA to NA] — Due to a small number of participants and events, data was not estimable. | NA [230 to NA] — Due to a small number of participants and events, data was not estimable.

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate (CBR) was defined as the number of participants documented to have a confirmed Complete Response (CR), Partial Response (PR), or Stable Disease (SD) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Participants who were not be able to be assessed for response were counted as non-responders.
Time Frame: Up to approximately 10 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Combination Regimen - Cohort 2: Participants with non-small cell lung cancer (NSCLC) who were naïve to treatment with immunotherapy, and had a tumor with no/low programmed cell death ligand 1 (PD-L1) expression were included in this cohort.
  Durvalumab - 1500 mg: Participants received durvalumab as an intravenous infusion every 4 weeks.
  Mocetinostat - Recommended Phase 2 Dose (70 mg): Participants received mocetinostat three times weekly as an oral capsule, at the dose recommended after Phase 1 (70 mg).
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
Number analyzed (Participants) | 5 | 4 | 9 | 15 | 3 | 21 | 13
Participants | 1 | 2 | 2 | 4 | 0 | 3 | 5

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from date of first study treatment to first Progressive Disease (PD) or death due to any cause in the absence of documented PD per RECIST v1.1
Time Frame: Randomization until progressive disease or death due to any cause (up to 42 months)
Population: Modified Intent-to-Treat Population (mITT) - The mITT Population was defined as all participants who received treatment with both mocetinostat and durvalumab on this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
Number analyzed (Participants) | 5 | 4 | 9 | 18 | 3 | 23 | 14
Months | 3 [1.88 to NA] — Due to a small number of participants and events, data was not estimable. | NA [NA to NA] — Due to a small number of participants and events, data was not estimable. | 2 [1.51 to 27.57] | 3 [2.01 to 5.86] | 4 [NA to NA] — Due to a small number of participants and events, data was not estimable. | 2 [1.94 to 14.57] | 3 [2.04 to 9.57]

7. Secondary Outcome: 1-Year Survival Rate
Time Frame: 1 year
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
Number analyzed (Participants) | 5 | 4 | 9 | 18 | 3 | 23 | 14
Proportion of participants | 0.40 [0.05 to 0.75] | 0.38 [0.01 to 0.81] | 0.53 [0.18 to 0.80] | 0.72 [0.41 to 0.89] | 1.00 [1.00 to 1.00] | 0.52 [0.31 to 0.70] | 0.50 [0.23 to 0.72]

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of study treatment to the date of death due to any cause.
Time Frame: From date of first study treatment until death due to any cause (up to 42 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
Number analyzed (Participants) | 5 | 4 | 9 | 18 | 3 | 23 | 14
Months | 7 [2.40 to 32.99] | 11 [7.17 to NA] — Due to a small number of participants and events, data was not estimable. | 16 [3.49 to 26.05] | NA [7.37 to NA] — Due to a small number of participants and events, data was not estimable. | NA [NA to NA] — Due to a small number of participants and events, data was not estimable. | 15 [7.73 to NA] — Due to a small number of participants and events, data was not estimable. | 14 [5.07 to 20.86]

9. Secondary Outcome: Concentration of Mocetinistat in Blood Plasma
Time Frame: Cycle 1 Day 1 pre-dose, 1, 3, and 7 hours post-dose, Cycle 1 Day 15 pre-dose and 1 hour post-dose, Cycle 2 Day 1 pre-dose and 1 hour post-dose, Cycle 3 Day 1 pre-dose and 1 hour post-dose and Cycle 7 Day 1 pre-dose (each cycle is 28 days)
Population: Pharmacokinetic Evaluable Population - The Pharmacokinetic (PK) Evaluable Population was defined as all patients who had PK concentration data collected for mocetinostat or durvalumab. Participants were combined for analysis of mocetinistat concentrations, as prespecified in the analysis shells, based on the actual dose of mocetinistat received in each phase of the study. Pharmacokinetic measures at 3 and 7 hours post dose on Cycle 1 Day 1 were only planned for Phase 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Phase 1: Mocetinostat 50 mg: The Phase 1 dose escalation established the recommended phase 2 dose (RP2D) of mocetinostat. Participants with advanced solid tumors were included in this Phase.
  Mocetinostat - 50 mg: Participants received mocetinostat three times weekly as an oral capsule.
  Durvalumab - 1500 mg: Participants received durvalumab as an intravenous infusion every 4 weeks.
- Phase 1: Mocetinostat 70 mg: The Phase 1 dose escalation established the recommended phase 2 dose (RP2D) of mocetinostat. Participants with advanced solid tumors were included in this Phase.
  Mocetinostat - 70 mg: Participants received mocetinostat three times weekly as an oral capsule.
  Durvalumab - 1500 mg: Participants received durvalumab as an intravenous infusion every 4 weeks.
- Phase 1: Mocetinostat 90 mg: The Phase 1 dose escalation established the recommended phase 2 dose (RP2D) of mocetinostat. Participants with advanced solid tumors were included in this Phase.
  Mocetinostat - 90 mg: Participants received mocetinostat three times weekly as an oral capsule.
  Durvalumab - 1500 mg: Participants received durvalumab as an intravenous infusion every 4 weeks.
- Phase 1: Mocetinostat 40 mg: One participant in Phase 1 was de-escalated to 40 mg of mocetinostat.
- Phase 2: Mocetinostat 70 mg: Participants in Phase 2 who received the recommended Phase 2 dose of 70 mg of mocetinostat.
- Phase 2: Mocetinostat 50 mg: Six participants in Phase 2 were de-escalated to 50 mg of mocetinostat.
Arm/Group | Phase 1: Mocetinostat 50 mg | Phase 1: Mocetinostat 70 mg | Phase 1: Mocetinostat 90 mg | Phase 1: Mocetinostat 40 mg | Phase 2: Mocetinostat 70 mg | Phase 2: Mocetinostat 50 mg
Number analyzed (Participants) | 9 | 7 | 11 | 1 | 63 | 6
ng/mL
  Cycle 1: Day 1 - pre-dose: number analyzed (Participants) | 4 | 3 | 6 | 0 | 59 | 0
  Cycle 1: Day 1 - pre-dose | NA (NA) — Geometric mean and corresponding coefficient of variation could not be estimated as none of the participants had an evaluable result (i.e. above LOQ). | 0.91 (83.20) | 1.02 (114.68) |  | 39.65 (175.97) |
  Cycle 1: Day 1 - 1 hour post-dose: number analyzed (Participants) | 4 | 3 | 6 | 0 | 59 | 0
  Cycle 1: Day 1 - 1 hour post-dose | 19.85 (441.16) | 106.61 (43.77) | 92.56 (143.96) |  | 12.19 (289.89) |
  Cycle 1: Day 1 - 3 hours post-dose: number analyzed (Participants) | 4 | 3 | 7 | 0 | 0 | 0
  Cycle 1: Day 1 - 3 hours post-dose | 33.53 (111.21) | 61.63 (24.78) | 55.27 (53.19) |  |  |
  Cycle 1: Day 1 - 7 hours post-dose: number analyzed (Participants) | 4 | 3 | 6 | 0 | 0 | 0
  Cycle 1: Day 1 - 7 hours post-dose | 15.75 (58.30) | 20.92 (27.20) | 33.89 (45.21) |  |  |
  Cycle 1: Day 15 - pre-dose: number analyzed (Participants) | 3 | 2 | 6 | 0 | 39 | 0
  Cycle 1: Day 15 - pre-dose | 5.36 (NA) — Geometric coefficient of variation could not be estimated as only one participant had an evaluable result (i.e. above LOQ). | 0.98 (95.06) | 3.84 (202.26) |  | 1.92 (127.96) |
  Cycle 1: Day 15 - 1 hour post-dose: number analyzed (Participants) | 3 | 2 | 4 | 0 | 37 | 0
  Cycle 1: Day 15 - 1 hour post-dose | 102.67 (7.17) | 22.30 (14646.88) | 18.32 (1297.79) |  | 10.86 (330.59) |
  Cycle 2: Day 1 - pre-dose: number analyzed (Participants) | 5 | 5 | 4 | 1 | 33 | 3
  Cycle 2: Day 1 - pre-dose | 0.72 (NA) — Geometric coefficient of variation could not be estimated as only one participant had an evaluable result (i.e. above LOQ). | 0.85 (NA) — Geometric coefficient of variation could not be estimated as only one participant had an evaluable result (i.e. above LOQ). | 1.22 (83.65) | NA (NA) — Geometric mean and corresponding coefficient of variation could not be estimated as none of the participants had an evaluable result (i.e. above LOQ). | 1.16 (91.63) | 0.68 (NA) — Geometric coefficient of variation could not be estimated as only one participant had an evaluable result (i.e. above LOQ).
  Cycle 2: Day 1 - 1 hour post-dose: number analyzed (Participants) | 4 | 5 | 5 | 1 | 35 | 3
  Cycle 2: Day 1 - 1 hour post-dose | 75.11 (25.53) | 49.30 (86.19) | 2.45 (83.60) | 0.72 (NA) — Geometric coefficient of variation could not be estimated as only one participant had an evaluable result (i.e. above LOQ). | 14.65 (396.22) | 105.00 (NA) — Geometric coefficient of variation could not be estimated as only one participant had an evaluable result (i.e. above LOQ).
  Cycle 3: Day 1 - pre-dose: number analyzed (Participants) | 6 | 1 | 0 | 1 | 18 | 3
  Cycle 3: Day 1 - pre-dose | 0.89 (44.73) | NA (NA) — Geometric mean and corresponding coefficient of variation could not be estimated as none of the participants had an evaluable result (i.e. above LOQ). |  | NA (NA) — Geometric mean and corresponding coefficient of variation could not be estimated as none of the participants had an evaluable result (i.e. above LOQ). | 4.08 (238.84) | 0.92 (40.65)
  Cycle 3: Day 1 - 1 hour post-dose: number analyzed (Participants) | 5 | 1 | 0 | 1 | 17 | 3
  Cycle 3: Day 1 - 1 hour post-dose | 22.73 (301.01) | 92.40 (NA) — Geometric coefficient of variation could not be estimated as only one participant had an evaluable result (i.e. above LOQ). |  | 0.73 (NA) — Geometric coefficient of variation could not be estimated as only one participant had an evaluable result (i.e. above LOQ). | 14.39 (319.34) | 25.12 (378.13)
  Cycle 7: Day 1 - pre-dose: number analyzed (Participants) | 1 | 1 | 1 | 0 | 8 | 1
  Cycle 7: Day 1 - pre-dose | NA (NA) — Geometric mean and corresponding coefficient of variation could not be estimated as none of the participants had an evaluable result (i.e. above LOQ). | 0.85 (NA) — Geometric coefficient of variation could not be estimated as only one participant had an evaluable result (i.e. above LOQ). | 1.35 (NA) — Geometric coefficient of variation could not be estimated as only one participant had an evaluable result (i.e. above LOQ). |  | 0.65 (35.19) | NA (NA) — Geometric mean and corresponding coefficient of variation could not be estimated as none of the participants had an evaluable result (i.e. above LOQ).

10. Secondary Outcome: Concentration of Durvalumab in Blood Plasma
Description: Plasma concentration of Durvalumab was evaluated. All participants received the same Durvalumab dose regardless of Mocetinistat dose group.
Time Frame: Cycle 1 Day 1 pre-dose + end of infusion, Cycle 1 Day 15 pre-mocetinostat dose, Cycle 2 Day 1 pre-dose, Cycle 3 Day 1 pre-dose, Cycle 4 Day 1 pre-dose + end of infusion, Cycle 7 Day 1 pre-dose + 90 days after participant's last dose (Up to max 133 weeks)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Durvalumab: Participants who received durvalumab during the study.
Arm/Group | Durvalumab
Number analyzed (Participants) | 76
ng/mL
  Cycle 1: Day 1 - pre-dose: number analyzed (Participants) | 70
  Cycle 1: Day 1 - pre-dose | 259.18 (334.86)
  Cycle 1: Day 1 - end of infusion: number analyzed (Participants) | 69
  Cycle 1: Day 1 - end of infusion | 385779.56 (36.49)
  Cycle 1: Day 15 - pre-Mocetinostat: number analyzed (Participants) | 49
  Cycle 1: Day 15 - pre-Mocetinostat | 102925.55 (40.05)
  Cycle 2: Day 1 - pre-dose: number analyzed (Participants) | 58
  Cycle 2: Day 1 - pre-dose | 44140.86 (130.83)
  Cycle 3: Day 1 - pre-dose: number analyzed (Participants) | 34
  Cycle 3: Day 1 - pre-dose | 72049.14 (91.22)
  Cycle 4: Day 1 - pre-dose: number analyzed (Participants) | 24
  Cycle 4: Day 1 - pre-dose | 101852.34 (89.01)
  Cycle 4: Day 1 - end of infusion: number analyzed (Participants) | 22
  Cycle 4: Day 1 - end of infusion | 365307.01 (81.59)
  Cycle 7: Day 1 - pre-dose: number analyzed (Participants) | 12
  Cycle 7: Day 1 - pre-dose | 130335.14 (70.34)
  90 days after last dose: number analyzed (Participants) | 24
  90 days after last dose | 12304.13 (501.74)

11. Secondary Outcome: Number of Participants With the Presence of Anti-Drug Antibody (ADA) in the Blood
Time Frame: Up to approximately 10 months
Population: ADA Evaluable Population - The ADA Evaluable Population was defined as all patients who received at least 1 dose of either durvalumab or mocetinostat for whom ADA results were available.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Combination Regimen - Cohort 1: Participants with non-small cell lung cancer (NSCLC) who were naïve to treatment with immunotherapy, and had a tumor with no/low programmed cell death ligand 1 (PD-L1) expression were included in this cohort.
  Durvalumab - 1500 mg: Participants received durvalumab as an intravenous infusion.
  Mocetinostat - Recommended Phase 2 Dose (70 mg): Participants received mocetinostat three times weekly as an oral capsule, at the dose recommended after Phase 1 (70 mg).
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
Number analyzed (Participants) | 1 | 4 | 9 | 17 | 3 | 22 | 15
Participants | 0 | 0 | 1 | 1 | 1 | 1 | 0

12. Secondary Outcome: Number of Participants With Tumor Expression of Programmed Cell Death Ligand 1 (PD-L1) at Baseline
Time Frame: Baseline
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
Number analyzed (Participants) | 5 | 4 | 9 | 18 | 3 | 23 | 14
Participants
  No/Low PD-L1 Expression | 0 | 0 | 0 | 17 | 0 | 6 | 9
  High PD-L1 Expression | 0 | 0 | 1 | 0 | 3 | 8 | 1
  Missing | 5 | 4 | 8 | 1 | 0 | 9 | 4

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are reported from the first day of study treatment until at least 28 days after last dose of study drug, and until resolution or stabilization of acute AEs (up to 125 weeks in Phase 1 and 92 weeks in Phase 2.) Serious adverse events (SAEs) are reported from the time of informed consent until 90 days after the last administration of mocetinostat or durvalumab (up to 133 weeks in Phase 1 and 101 weeks in Phase 2.)
Groups:
- Phase 1: Dose Escalation - 50 mg; Phase 1: Dose Escalation - 70 mg; Phase 1: Dose Escalation - 90 mg: The Phase 1 dose escalation established the recommended phase 2 dose (RP2D) of mocetinostat. Participants with advanced solid tumors were included in this phase.
  Mocetinostat: Participants received mocetinostat three times weekly as an oral capsule.
  Durvalumab - 1500 mg: Participants received durvalumab as an intravenous infusion every 4 weeks.
Arm/Group | Phase 1: Dose Escalation - 50 mg | Phase 1: Dose Escalation - 70 mg | Phase 1: Dose Escalation - 90 mg | Phase 2: Combination Regimen - Cohort 1 | Phase 2: Combination Regimen - Cohort 2 | Phase 2: Combination Regimen - Cohort 3 | Phase 2: Combination Regimen - Cohort 4
All-Cause Mortality (participants affected / at risk) | 5/5 | 2/4 | 9/11 | 5/18 | 0/3 | 14/23 | 12/19
Serious Adverse Events (participants affected / at risk) | 4/5 | 1/4 | 4/11 | 6/18 | 2/3 | 5/23 | 11/19
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 10/11 | 18/18 | 3/3 | 23/23 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Dose Escalation - 50 mg (N=5) | Phase 1: Dose Escalation - 70 mg (N=4) | Phase 1: Dose Escalation - 90 mg (N=11) | Phase 2: Combination Regimen - Cohort 1 (N=18) | Phase 2: Combination Regimen - Cohort 2 (N=3) | Phase 2: Combination Regimen - Cohort 3 (N=23) | Phase 2: Combination Regimen - Cohort 4 (N=19)
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 2 | 4
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis adenovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0 | 0 | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Dose Escalation - 50 mg (N=5) | Phase 1: Dose Escalation - 70 mg (N=4) | Phase 1: Dose Escalation - 90 mg (N=11) | Phase 2: Combination Regimen - Cohort 1 (N=18) | Phase 2: Combination Regimen - Cohort 2 (N=3) | Phase 2: Combination Regimen - Cohort 3 (N=23) | Phase 2: Combination Regimen - Cohort 4 (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 3 | 1 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 3 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Episcleritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 9 | 7 | 3 | 10 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 4 | 9 | 1 | 11 | 9
Vomiting (Gastrointestinal disorders) | 4 | 1 | 8 | 4 | 1 | 6 | 5
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 3 | 1 | 6 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorectal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal wall thickening (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal dilatation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 7 | 11 | 3 | 14 | 8
Oedema peripheral (General disorders) | 0 | 0 | 2 | 1 | 0 | 3 | 3
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 2
Asthenia (General disorders) | 1 | 0 | 1 | 2 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 2
Chills (General disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 3
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Early satiety (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site discharge (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 4 | 0 | 3 | 2
Cystitis (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stoma site irritation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 3 | 3 | 0 | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 4 | 7 | 1 | 7 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0 | 4 | 1 | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 2 | 0 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 4 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 1 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 2 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 4 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 2 | 0 | 4 | 1
Headache (Nervous system disorders) | 2 | 0 | 1 | 1 | 0 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device occlusion (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 6 | 0 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 4 | 0 | 4 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Umbilical erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2 | 3 | 0 | 0 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was discontinued early because the Sponsor de-prioritized development of mocetinostat. The decision to stop was not due to any patient safety issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can not disclose, discuss, or publish study results until final manuscript has been published.

DOCUMENTS (2):
  • Study Protocol (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT02805660/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT02805660/SAP_001.pdf